CLINICAL TRIAL: NCT02393001
Title: Analysis of Skin Lesions for Melanoma Presence by Volatile Spectroscopy Techniques
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201400739
Record Dates: First submitted 2015-03-09; First posted 2015-03-19 (Estimated); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Melanoma
Keywords: skin cancer; suspicious lesion; skin biopsy; noninvasive; screening
MeSH Terms: conditions — Melanoma; Skin Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Dermatology patients: Patients seen in the dermatology clinic with suspicious skin lesion to be biopsied will have 4 skin swabs, 2 of the skin lesion and 2 of an area of unafflicted skin.
  Interventions: Other: Dermatology patients

INTERVENTIONS:
Other: Dermatology patients — Cleanse an area of unafflicted (control) skin with a cotton 2 x 2 dampened with saline.
Other: Dermatology patients — Cleanse a suspicious lesion (potential melanoma) with a saline cotton swab.
Other: Dermatology patients — This intervention follows the standard of care for patients with a suspicious skin lesion (potential melanoma) the physician plans to biopsy. The alcohol swab used to prep the site will be stored for testing rather than discarded.
Other: Dermatology patients — Cleanse an area of unafflicted (control) skin with an alcohol swab.

SUMMARY:
The purpose of this research study is to determine if a very sensitive chemistry lab analyzer can be used to smell a skin cancer (like melanoma) similar to some dogs.

DETAILED DESCRIPTION:
Types of skin cancer, like melanoma, are likely to spread and are becoming increasingly common. At this time, healthcare providers look at patient's skin and remove a sample of suspicious areas of the skin (biopsy) to test for cancer.

This research study will inspect cotton and cloth swabs of normal skin and suspicious areas of the skin that are going to be biopsied just before the biopsy. The swabs will be looked at with a very sensitive chemistry lab analyzer to see if the lab analyzer can confirm conventional lab test findings.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Seen at the dermatology clinic & determined to need a skin biopsy of a suspicious lesion

Exclusion Criteria:

* < 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients seen in the dermatology clinic with suspicious skin lesion to be biopsied will have 4 skin swabs, 2 of the skin lesion and 2 of an area of unafflicted skin
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2015-05; Primary Completion 2017-09-30 (Actual); Study Completion 2017-10-03 (Actual)

PRIMARY OUTCOMES:
Compare the off line spectral analyses of saline and alcohol skin swabs of normal control, melanoma negative and melanoma positive skin biopsies. | 1 day
  Determine if the melanomas have unique identifying spectra that might be applied to noninvasive melanoma skin cancer screening in lieu of taking a biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Nikolaus Gravenstein, MD, Principal Investigator — The Jerome H. Modell, MD, Professor of Anesthesiology
Locations (1):
- UF Health, Gainesville, Florida, United States